CLINICAL TRIAL: NCT03830333
Title: A Phase 3, Multicenter, Double-blind, Randomized, Active-controlled Clinical Study to Evaluate the Efficacy and Safety of Ceftolozane/Tazobactam (MK-7625A) Plus Metronidazole Versus Meropenem in Chinese Participants With Complicated Intra-abdominal Infection
Brief Title: Ceftolozane/Tazobactam (MK-7625A) Plus Metronidazole Versus Meropenem for Participants With Complicated Intra-abdominal Infection (MK-7625A-015)
Acronym: 7625ACNPhase3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7625A-015; MK-7625A-015 (Other: Merck)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Complicated Intra-abdominal Infections
MeSH Terms: interventions — ceftolozane, tazobactam drug combination; Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ceftolozane/Tazobactam + Metronidazole (Experimental): Participants receive ceftolozane/tazobactam 1500 mg (ceftolozane 1000 mg + tazobactam 500 mg) plus metronidazole 500 mg administered as an intravenous (IV) infusion every 8 hours for 4 to 14 days (per protocol, ceftolozane/tazobactam may be adjusted to 500 mg/250 mg if creatinine clearance [CrCL] is 30 to ≤50 mL/min)
  Interventions: Drug: Ceftolozane/Tazobactam; Drug: Metronidazole
- Meropenem + Placebo (Active Comparator): Participants receive meropenem 1000 mg plus saline administered as an IV infusion every 8 hours for 4 to 14 days (per protocol, meropenem may be adjusted to every 12 hours if CrCL was 30 to ≤50 mL/min).
  Interventions: Drug: Meropenem; Drug: Placebo

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam — Ceftolozane 1000 mg / tazobactam 500 mg by IV infusion every 8 hours for 4 to 14 days. Participants with CrCL of 30 to ≤ 50 mL/min will receive ceftolozane 500 mg / tazobactam 250 mg.
  Other Names: MK-7625A
  Arms: Ceftolozane/Tazobactam + Metronidazole
Drug: Metronidazole — Metronidazole 500 mg by IV infusion every 8 hours for 4 to 14 days.
  Arms: Ceftolozane/Tazobactam + Metronidazole
Drug: Meropenem — Meropenem 1000 mg by IV infusion every 8 hours for 4 to 14 days. Participants with CrCL of 30 to ≤ 50 mL/min will receive IV infusion every 12 hours.
  Arms: Meropenem + Placebo
Drug: Placebo — Saline by IV infusion every 8 hours for 4 to 14 days.
  Arms: Meropenem + Placebo

SUMMARY:
This study aims to evaluate the efficacy of ceftolozane/tazobactam (MK-7625A) plus metronidazole versus meropenem in adults diagnosed with complicated intra-abdominal infection (cIAI). The primary hypothesis is ceftolozane/tazobactam plus metronidazole is non-inferior to meropenem, as measured by the clinical response rate at the Test-of Cure (TOC) visit in the Clinically Evaluable (CE) population.

ELIGIBILITY:
Inclusion Criteria:

* Must have one of the following diagnoses in which there is evidence of bacterial intraperitoneal infection: Cholecystitis (including gangrenous cholecystitis) with rupture, perforation, or progression of the infection beyond the gallbladder wall; Acute gastric or small intestine including duodenal perforation, only if operated on > 24 hours after perforation occurs; Traumatic perforation of the intestine (including colon), only if operated on > 12 hours after perforation occurs; Appendiceal perforation or peri-appendiceal abscess; Diverticular disease with perforation or abscess; Peritonitis due to other perforated viscus or following a prior operative procedure; Intra-abdominal abscess (including liver or spleen).
* Evidence of systemic infection
* Requires surgical intervention (e.g., laparotomy, laparoscopic surgery, or percutaneous draining of an abscess) within 24 hours of (before or after) the first dose of study drug
* If participant is to be enrolled preoperatively, the participant should have radiographic evidence of gastric or bowel perforation or intra-abdominal abscess or other radiographic evidence for cIAI
* Participants who failed prior antibacterial treatment for the current cIAI can be enrolled but must: (a) have a positive culture (from an intra-abdominal site or blood sample) and (b) require surgical intervention.
* Is a Chinese participant, defined as a person of Chinese descent. A potential participant who is of ex-China descent (e.g. Western European) descent living in China will be excluded
* Male agrees to use contraception during the treatment period, and for at least 30 days after the last dose of study medication, and refrain from donating sperm during this period
* Female is not pregnant or breastfeeding; is not a woman of childbearing potential (WOCBP); or if WOCBP agrees to use a contraceptive method that is highly effective, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle during the treatment period, and for at least 30 days after the last dose of study medication; or must have a negative highly sensitive pregnancy test (serum) within 48 hours before the first dose of study intervention.

Exclusion Criteria:

* Has any of the following diagnoses: simple appendicitis; abdominal wall abscess; small bowel obstruction or ischemic bowel disease without perforation; spontaneous (primary) bacterial peritonitis associated with cirrhosis and chronic ascites; or pelvic infections
* Has any of the following diseases: acute suppurative cholangitis; infected necrotizing pancreatitis; pancreatic abscess
* Has complicated intra-abdominal infection managed by staged abdominal repair (STAR), open abdomen technique (i.e. fascia not closed) including temporary closure of the abdomen, or any situation where infection source control was not likely to be achieved
* Has abscess that is confirmed on imaging test but has not been or cannot be managed by surgical intervention including drainage
* Is expected to be cured by only surgical intervention (e.g., drainage) without use of systemic antibiotic therapy
* Has the following underlying conditions or the following serious conditions: considered unlikely to survive during the study period (predicted life expectancy is < 4 weeks after randomization); organic brain or spinal cord disease; any rapidly-progressing disease or immediately life-threatening illness (including respiratory failure and septic shock); an immunocompromising condition
* Has a history of any hypersensitivity or allergic reaction to any beta-lactam, antibacterials, including cephalosporins, carbapenems, penicillins, or tazobactam, or metronidazole, or nitroimidazole derivatives; or if a skin test is required by local clinical regulations, has a positive skin test result if no prior history of allergic reaction to beta-lactam antibacterials
* A WOCBP who has a positive serum pregnancy test within 24 hours before the first dose of study intervention
* Used systemic antibiotic therapy with known coverage of pathogens that cause IAI for more than 24 hours during the previous 72 hours prior to the first dose of study drug, unless there is a documented treatment failure with such therapy
* For participants that are enrolled postoperatively, more than 1 dose of an active non-study antibacterial regimen administered postoperatively. For participants enrolled preoperatively, no postoperative non-study antibacterial therapy is allowed
* Participants who need additional non-study systemic antibacterial therapy with gram-negative activity in addition to study drug therapy; drugs with only gram-positive activity (eg, IV vancomycin, teicoplanin, linezolid and daptomycin) are allowed
* Anticipates treatment with traditional Chinese medicine or herbal medicine during study period
* Has received disulfiram, valproic acid or divalproex sodium within 14 days before the proposed first day of study drug or who are currently receiving probenecid
* Is currently participating in, or has participated in, any other clinical study involving the administration of investigational or experimental medication (not licensed by regulatory agencies) at the time of the presentation or during the previous 90 days prior to screening or is anticipated to participate in such a clinical study during the course of this study
* Has participated in a ceftolozane/tazobactam clinical study at any time in the past
* Has severe impairment of renal function (CrCL <30 mL/min) or requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- China (25):
  - Anhui Provincial Hospital ( Site 0033), Hefei, Anhui
  - Navy General Hospital ( Site 0009), Beijing, Beijing Municipality
  - Peking University Third Hospital ( Site 0002), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0026), Guangzhou, Guangdong
  - Hainan General Hospital ( Site 0042), Haikou, Hainan
  - Baotou Central Hospital ( Site 0013), Baotou, Inner Mongolia
  - The First People's Hospital of Changzhou ( Site 0054), Changzhou, Jiangsu
  - Wuxi No.2 People's Hospital ( Site 0050), Wuxi, Jiangsu
  - Wuxi People's Hospital ( Site 0020), Wuxi, Jiangsu
  - Subei People's Hospital ( Site 0046), Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University ( Site 0049), Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 0029), Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University ( Site 0053), Nanchang, Jiangxi
  - The Second Hospital of Jilin University ( Site 0048), Changchun, Jilin
  - Liaocheng People s hospital ( Site 0014), Liaocheng, Shandong
  - Zhongshan Hospital of Fudan University ( Site 0001), Shanghai, Shanghai Municipality
  - Shanghai General Hospital ( Site 0016), Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District ( Site 0052), Shanghai, Shanghai Municipality
  - Tianjin People's Hospital ( Site 0040), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University ( Site 0034), Ürümqi, Xinjiang
  - The First Hospital of Kunming ( Site 0041), Kunming, Yunnan
  - Taizhou Hospital of Zhejiang Province ( Site 0035), Taizhou, Zhejiang
  - The 2nd Affiliated Hospital of Wenzhou Medical University ( Site 0051), Wenzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0015), Wenzhou, Zhejiang
  - Southern Medical University Nanfang Hospital ( Site 0055), Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sun Y, Fan J, Chen G, Chen X, Du X, Wang Y, Wang H, Sun F, Johnson MG, Bensaci M, Huntington JA, Bruno CJ. A phase III, multicenter, double-blind, randomized clinical trial to evaluate the efficacy and safety of ceftolozane/tazobactam plus metronidazole versus meropenem in Chinese participants with complicated intra-abdominal infections. Int J Infect Dis. 2022 Oct;123:157-165. doi: 10.1016/j.ijid.2022.08.003. Epub 2022 Aug 17. PMID 35987467
- [Derived] Li Z, Kang Y, Gao H, Zhao Y, Luo D, Wang D, Zhang X, Yu J, Chu G, Cao J, Wang F, Zhao X, Jensen E, Lin G, Chen G. Pooled data from phase 3 clinical trials comparing the clinical activity of ceftolozane/tazobactam versus meropenem for the treatment of complicated intra-abdominal infections. Infect Dis (Lond). 2026 Jan;58(1):40-51. doi: 10.1080/23744235.2025.2544828. Epub 2025 Sep 6. PMID 40913503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with complicated intra-abdominal infection (cIAI) were recruited at 21 study sites in China. Participants with severe impairment of renal function (estimated creatinine clearance [CrCL] <30 mL/min) were excluded.
Groups:
- Ceftolozane/Tazobactam + Metronidazole: Participants received ceftolozane/tazobactam 1500 mg (ceftolozane 1000 mg + tazobactam 500 mg) plus metronidazole 500 mg administered as an intravenous (IV) infusion every 8 hours for 4 to 14 days (per protocol, ceftolozane/tazobactam could be adjusted to 500 mg/250 mg if CrCL was 30 to ≤50 mL/min).
- Meropenem + Placebo: Participants received meropenem 1000 mg plus saline administered as an IV infusion every 8 hours for 4 to 14 days (per protocol, meropenem could be adjusted to every 12 hours if CrCL was 30 to ≤50 mL/min).
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Started | 134 | 134
Clinically Evaluable Population | 105 | 116
Completed | 126 | 130
Not Completed | 8 | 4
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Discontinuations associated with failure to return for follow-up assessments due to COVID-19 | 3 | 2

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population consisted of all randomized participants. Participants in the ITT population were analyzed based on the treatment they were randomized to, irrespective of what they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo | Total
Number analyzed (Participants) | 134 | 134 | 268
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (16.2) | 51.1 (15.7) | 49.3 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 79 | 85 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 134 | 134 | 268
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 134 | 134 | 268
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Primary Site of Infection [Count of Participants; unit: Participants] — Primary site of infection consisted of bowel (small or large) and other site of infection. Participants with appendix, stomach, or duodenum as the anatomic site of infection, were stratified to the "other site" group.
  Participants
    Bowel (small or large) | 5 | 8 | 13
    Other site of infection | 129 | 126 | 255

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response (Clinical Cure or Clinical Failure) at Test of Cure (TOC) Visit: Clinically Evaluable (CE) Population
Description: Clinical response was classified as "cure" or "failure". Clinical cure (favorable) was defined as complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required for the index infection. Clinical failure (unfavorable) was defined as death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care. The percentage of participants with clinical response of clinical cure or clinical failure at TOC was summarized.
Time Frame: Up to approximately Day 30
Population: All participants of the CE population who met the protocol definition of cIAI, had no significant protocol deviations, received the minimum duration of randomized IV study therapy, and had an efficacy assessment of cure or failure at the TOC visit were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 105 | 116
Percentage of Participants
  Clinical Cure (favorable) | 95.2 | 93.1
  Clinical Failure (unfavorable) | 4.8 | 6.9
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Difference in percentage was based on Miettinen and Nurminen method with the Cochran-Mantel-Haenszel (CMH) weighting stratified by anatomic site of infection (bowel [small or large] versus other site of cIAI); Test type: Non-Inferiority — Ceftolozane/tazobactam + metronidazole is concluded to be non-inferior to meropenem + placebo if the lower bound of the 95% CI for the treatment difference in percent response is above -12.5 percentage points; Difference in percentages = 2.1, 95% CI 2-sided [-4.7 to 8.8]

2. Secondary Outcome: Percentage of Participants With Clinical Response (Clinical Cure, Clinical Failure, or Indeterminate) at TOC Visit: Intent to Treat (ITT) Population
Description: Clinical response was classified as "cure", "failure", or "indeterminate". Clinical cure (favorable) was defined as complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required for the index infection. Clinical failure (unfavorable) was defined as death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care. Indeterminate (unfavorable) was defined as participants for whom study data were not available for evaluation of efficacy for any reason. The percentage of participants with clinical response of clinical cure, clinical failure, or indeterminate at TOC was summarized.
Time Frame: Up to approximately Day 30
Population: The ITT population consisted of all randomized participants. Participants in the ITT population were analyzed based on the treatment they were randomized to, irrespective of what they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 134 | 134
Percentage of Participants
  Clinical Cure (favorable) | 85.1 | 89.6
  Clinical Failure (unfavorable) | 14.2 | 9.7
  Indeterminate (unfavorable) | 0.7 | 0.7
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Difference in percentage was based on Miettinen and Nurminen method with the CMH weighting stratified by anatomic site of infection (bowel [small or large] versus other site of cIAI); Test type: Other; Difference in percentages = -4.4, 95% CI 2-sided [-12.6 to 3.7]

3. Secondary Outcome: Percentage of Participants With Clinical Response (Clinical Cure or Clinical Failure) at End of Therapy (EOT) Visit: CE Population
Description: Clinical response was classified as "cure" or "failure". Clinical cure (favorable) was defined as complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required for the index infection. Clinical failure (unfavorable) was defined as death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care. The percentage of participants with clinical response of clinical cure or clinical failure at EOT was summarized.
Time Frame: Up to approximately Day 15
Population: All participants of the CE population who met the protocol definition of cIAI, had no significant protocol deviations, received the minimum duration of randomized IV study therapy, and had an efficacy assessment of cure or failure at the EOT visit were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 105 | 116
Percentage of Participants
  Clinical Cure (favorable) | 98.1 | 96.6
  Clinical Failure (unfavorable) | 1.9 | 3.4
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference in percentages = 1.4, 95% CI 2-sided [-3.8 to 6.7]

4. Secondary Outcome: Percentage of Participants With Clinical Response (Clinical Cure, Clinical Failure, or Indeterminate) at EOT Visit: ITT Population
Description: Clinical response was classified as "cure", "failure", or "indeterminate". Clinical cure (favorable) was defined as complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure is required for the index infection. Clinical failure (unfavorable) was defined as death related to IAI at any time point; persisting or recurrent infection within the abdomen requiring additional intervention to cure; need for treatment with additional antibiotics for ongoing IAI symptoms; or post-surgical wound infection that requires additional antimicrobial therapy and/or non-routing wound care. Indeterminate (unfavorable) was defined as participants for whom study data are not available for evaluation of efficacy for any reason. The percentage of participants with clinical response of clinical cure, clinical failure, or indeterminate at EOT was summarized.
Time Frame: Up to approximately Day 15
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 134 | 134
Percentage of Participants
  Clinical Cure (favorable) | 92.5 | 94.0
  Clinical Failure (unfavorable) | 7.5 | 4.5
  Indeterminate (unfavorable) | 0.0 | 1.5
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Difference in percentages = -1.5, 95% CI 2-sided [-8.0 to 4.8]

5. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response of Eradication or Presumed Eradication at TOC Visit: Expanded Microbiologically Evaluable (EME) Population
Description: An overall microbiological response was determined by the Sponsor for each participant based on individual microbiological responses for each baseline bacterial pathogen. A favorable individual microbiological response was eradication (absence of the baseline bacterial pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a participant who is assessed as a clinical cure). In order for the participant to have a favorable overall microbiological response, each individual baseline bacterial pathogen must have had a favorable microbiological outcome. The percentage of participants with a favorable per-participant microbiological response of eradication or presumed eradication was reported for the TOC visit.
Time Frame: Up to approximately Day 30
Population: The EME population consisted of all randomized participants who had cIAI as evidenced by identification of at least 1 baseline intra-abdominal pathogen, regardless of susceptibility to study drug and met all CE population criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 54 | 73
Percentage of Participants | 94.4 | 93.2
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Difference in percentage based on Miettinen and Nurminen method with the CMH weighting stratified by anatomic site of infection (bowel [small or large] versus other site of cIAI); Test type: Other; Difference in percentages = 1.2, 95% CI 2-sided [-9.2 to 10.4]

6. Secondary Outcome: Percentage of Participants With Favorable Microbiological Response of Eradication or Presumed Eradication, by Pathogen, at the TOC Visit: EME Population
Description: A microbiological response was determined for each bacterial pathogen isolated at baseline by the Sponsor. Favorable microbiological responses included eradication (absence of the baseline bacterial pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a participant who is assessed as a clinical cure). The percentage of participants with a favorable microbiological response of eradication or presumed eradication was reported per pathogen for the TOC visit.
Time Frame: Up to approximately Day 30
Population: The EME population consisted of all randomized participants with data available who had cIAI as evidenced by identification of at least 1 baseline intra-abdominal pathogen, regardless of susceptibility to study drug and met all CE population criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 54 | 73
Percentage of Participants
  Gram-negative aerobes: number analyzed (Participants) | 50 | 60
  Gram-negative aerobes | 94.0 | 95.0
  All Enterobacteriaceae: number analyzed (Participants) | 48 | 60
  All Enterobacteriaceae | 93.8 | 95.0
  Citrobacter freundii complex: number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex | 100.0 |
  Citrobacter koseri: number analyzed (Participants) | 1 | 0
  Citrobacter koseri | 100.0 |
  Enterobacter aerogenes: number analyzed (Participants) | 1 | 0
  Enterobacter aerogenes | 100.0 |
  Enterobacter cloacae complex: number analyzed (Participants) | 2 | 0
  Enterobacter cloacae complex | 100.0 |
  Other Enterobacter spp.: number analyzed (Participants) | 0 | 2
  Other Enterobacter spp. |  | 100.0
  Escherichia coli: number analyzed (Participants) | 32 | 46
  Escherichia coli | 93.8 | 95.7
  Klebsiella oxytoca: number analyzed (Participants) | 0 | 3
  Klebsiella oxytoca |  | 100.0
  Klebsiella pneumoniae: number analyzed (Participants) | 11 | 11
  Klebsiella pneumoniae | 100.0 | 90.9
  Morganella morganii: number analyzed (Participants) | 0 | 1
  Morganella morganii |  | 100.0
  Proteus mirabilis: number analyzed (Participants) | 2 | 0
  Proteus mirabilis | 50.0 |
  Aeromonas hydrophila: number analyzed (Participants) | 1 | 0
  Aeromonas hydrophila | 100.0 |
  Pseudomonas aeruginosa: number analyzed (Participants) | 4 | 1
  Pseudomonas aeruginosa | 75.0 | 100.0
  Gram-positive aerobes: number analyzed (Participants) | 10 | 17
  Gram-positive aerobes | 80.0 | 88.2
  Gram-negative anaerobes: number analyzed (Participants) | 0 | 1
  Gram-negative anaerobes |  | 100.0
  Gram-positive anaerobes: number analyzed (Participants) | 1 | 1
  Gram-positive anaerobes | 100.0 | 100.0
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Gram-negative aerobes comparison: Based on unstratified Miettinen and Nurminen method; Test type: Other — Difference in percentage was based on unstratified Miettinen and Nurminen method. Confidence Interval is displayed only when there are at least 4 participants in at least one treatment group; Difference in percentages = -1.0, 95% CI 2-sided [-11.9 to 8.7]
Statistical Analysis 2: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; All enterobacteriaceae comparison: Based on unstratified Miettinen and Nurminen method; Test type: Other — [test comment as in outcome 6, analysis 1]; Difference in percentages = -1.2, 95% CI 2-sided [-12.5 to 8.5]
Statistical Analysis 3: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Gram-positive aerobes comparison: Based on unstratified Miettinen and Nurminen method; Test type: Other — [test comment as in outcome 6, analysis 1]; Difference in percentages = -8.2, 95% CI 2-sided [-42.2 to 20.0]

7. Secondary Outcome: Percentage of Participants Who Experienced 1 or More Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. The percentage of participants who experienced 1 or more AEs were summarized.
Time Frame: Up to approximately Day 30
Population: The All Participants as Treated (APaT) population was used for the analysis of safety data in this study. The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 134 | 134
Percentage of Participants | 50.0 | 50.7
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Difference in percentage was based on Miettinen & Nurminen method; Test type: Other; Difference in Percentages = -0.7, 95% CI 2-sided [-12.6 to 11.2]

8. Secondary Outcome: Percentage of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. The percentage of participants who had study drug discontinued during the study due to an AE was summarized.
Time Frame: Up to Day 14
Population: The APaT population was used for the analysis of safety data in this study. The APaT population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
Number analyzed (Participants) | 134 | 134
Percentage of Participants | 2.2 | 2.2
Statistical Analysis 1: Comparison: Ceftolozane/Tazobactam + Metronidazole vs Meropenem + Placebo; Difference in percentage was based on Miettinen & Nurminen method; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-4.4 to 4.4]

ADVERSE EVENTS:
Time Frame: Up to approximately Day 30
Description: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Ceftolozane/Tazobactam + Metronidazole | Meropenem + Placebo
All-Cause Mortality (participants affected / at risk) | 0/134 | 1/134
Serious Adverse Events (participants affected / at risk) | 7/134 | 7/134
Other Adverse Events (participants affected / at risk) | 28/134 | 33/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam + Metronidazole (N=134) | Meropenem + Placebo (N=134)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 2 (2) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam + Metronidazole (N=134) | Meropenem + Placebo (N=134)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 11 (12)
Pyrexia (General disorders) | 9 (11) | 14 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03830333/Prot_SAP_000.pdf